CLINICAL TRIAL: NCT03435679
Title: One-stage Versus Two-stage Revision of the Infected Knee Arthroplasty. a Randomized Controlled Multicenter Trial.
Brief Title: One-stage Versus Two-stage Revision of the Infected Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Martin Lindberg-Larsen, Orthopaedic Surgeon, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLL_02_2018
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Periprosthetic Knee Infection
Keywords: infection; knee arthroplasty; surgical treatment; one-stage; two-stage; outcome
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- one-stage (Experimental): one-stage surgical treatment of the infected knee arthroplasty
  Interventions: Procedure: one-stage
- two-stage (Active Comparator): two-stage surgical treatment of the infected knee arthroplasty with a interim period of 8-10 weeks between stages
  Interventions: Procedure: two-stage

INTERVENTIONS:
Procedure: one-stage — one-stage surgery
  Arms: one-stage
Procedure: two-stage — two-stage surgery
  Arms: two-stage

SUMMARY:
This study investigates functional outcome and safety after one-stage versus two-stage revision of the infected knee arthroplasty.

Half of participants are treated with a one-stage surgical procedure, while the other half is treated with a two-stage procedure.

The investigators hypothesize that the functional outcome and quality of life of the participants is superior after one-stage surgery compared to two-stage surgery.

DETAILED DESCRIPTION:
A two-stage approach is the standard surgical procedure in the treatment of the chronically infected knee arthroplasty, but promising results have been reported after a one-stage approach from single-centre studies.

The potential benefits for the patients treated with a one-stage approach are many as they only have to go through surgery and rehabilitation once with shorter total length of hospital stay. However, no randomized controlled trials comparing outcome after the procedures have been performed so far.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of periprosthetic knee infection
* > 6 weeks from previous knee arthoplasty procedure (primary or total revision procedure)
* Speak and understand Danish and have given informed consent

Exclusion Criteria:

* Soft tissue problems requiring plastic surgery
* major bone loss requiring mega/tumor-prosthesis
* acute surgery due to sepsis
* malignant disease with less than 2 years life expectancy
* re-infection with previous two-stage procedure
* bilateral knee infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (AUC) | preoperatively 6 weeks, 3, 6, 9, 12 months postoperatively.
  Area Under Curve for Oxford Knee Score

SECONDARY OUTCOMES:
Oxford Knee Score (AUC) | preoperatively, 6 weeks, 3, 6, 9, 12, 18 and 24 months postoperatively.
  Area Under Curve for Oxford Knee Score
EQ-5D-5L | preoperatively, 6 weeks, 3, 6, 9, 12, 18 and 24 months postoperatively.
  Quality of life questionnaire
Re-revision rate | 2 year postoperatively
  re-revisions due to infection and other causes
mortality | 90 days postoperatively and 1 and 2 year postoperatively
  postoperative mortality
readmission rate | 90 days postoperatively
  postoperative readmission rate
Range of Motion | 2 years postoperatively
  Range of motion of the infected/operated knee

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lindberg-Larsen, Principal Investigator — Martin Lindberg-Larsen
Locations (9):
- Denmark (9):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Horsens Hospital, Horsens
  - Næstved Hospital, Næstved
  - Odense Universitets Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No
According to local interpretation of GDPR. Blinded data can be provided upon request.

REFERENCES:
- [Background] Lindberg-Larsen M, Jorgensen CC, Bagger J, Schroder HM, Kehlet H. Revision of infected knee arthroplasties in Denmark. Acta Orthop. 2016 Aug;87(4):333-8. doi: 10.3109/17453674.2016.1148453. Epub 2016 Feb 22. PMID 26900908
- [Background] Lindberg-Larsen M, Pitter FT, Voldstedlund M, Schroder HM, Bagger J. Microbiological diagnosis in revision of infected knee arthroplasties in Denmark. Infect Dis (Lond). 2017 Nov-Dec;49(11-12):824-830. doi: 10.1080/23744235.2017.1350878. Epub 2017 Jul 8. PMID 28691647
- [Background] Masters JP, Smith NA, Foguet P, Reed M, Parsons H, Sprowson AP. A systematic review of the evidence for single stage and two stage revision of infected knee replacement. BMC Musculoskelet Disord. 2013 Jul 29;14:222. doi: 10.1186/1471-2474-14-222. PMID 23895421
- [Background] Haddad FS, Sukeik M, Alazzawi S. Is single-stage revision according to a strict protocol effective in treatment of chronic knee arthroplasty infections? Clin Orthop Relat Res. 2015 Jan;473(1):8-14. doi: 10.1007/s11999-014-3721-8. PMID 24923669
- [Background] Singer J, Merz A, Frommelt L, Fink B. High rate of infection control with one-stage revision of septic knee prostheses excluding MRSA and MRSE. Clin Orthop Relat Res. 2012 May;470(5):1461-71. doi: 10.1007/s11999-011-2174-6. Epub 2011 Nov 12. PMID 22081299
- [Background] Baker P, Petheram TG, Kurtz S, Konttinen YT, Gregg P, Deehan D. Patient reported outcome measures after revision of the infected TKR: comparison of single versus two-stage revision. Knee Surg Sports Traumatol Arthrosc. 2013 Dec;21(12):2713-20. doi: 10.1007/s00167-012-2090-7. Epub 2012 Jun 13. PMID 22692517
- [Background] Massin P, Delory T, Lhotellier L, Pasquier G, Roche O, Cazenave A, Estellat C, Jenny JY. Infection recurrence factors in one- and two-stage total knee prosthesis exchanges. Knee Surg Sports Traumatol Arthrosc. 2016 Oct;24(10):3131-3139. doi: 10.1007/s00167-015-3884-1. Epub 2015 Nov 26. PMID 26611899
- [Derived] Lindberg-Larsen M, Odgaard A, Fredborg C, Schroder HM; One-stage vs Two-stage Collaboration Group. One-stage versus two-stage revision of the infected knee arthroplasty - a randomized multicenter clinical trial study protocol. BMC Musculoskelet Disord. 2021 Feb 12;22(1):175. doi: 10.1186/s12891-021-04044-8. PMID 33579256